CLINICAL TRIAL: NCT03989596
Title: Hypofractionated Radiotherapy With Hyperthermia in Unresectable or Marginally Resectable Soft Tissue Sarcomas
Acronym: SINDIR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SINDIR1
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2020-12

CONDITIONS: Sarcoma; Alveolar Soft Part Sarcoma; Clear Cell Sarcoma; Malignant Peripheral Nerve Sheath Tumors; Myxoid Liposarcoma; Liposarcoma, Dedifferentiated; Synovial Sarcoma; Leiomyosarcoma; Undifferentiated Pleomorphic Sarcoma; Fibrosarcoma; Pleomorphic Rhabdomyosarcoma
Keywords: Dose Hypofractionation; Neoadjuvant Therapy; Sarcoma; Hyperthermia; Dose Fractionation
MeSH Terms: conditions — Sarcoma; Sarcoma, Alveolar Soft Part; Sarcoma, Clear Cell; Neurofibrosarcoma; Liposarcoma, Myxoid; Liposarcoma; Sarcoma, Synovial; Leiomyosarcoma; Histiocytoma, Malignant Fibrous; Fibrosarcoma; Hyperthermia | interventions — Radiation Dose Hypofractionation; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy with hyperthermia (Experimental): 10x 3.25 Gy + hyperthermia + surgery or radiotherapy boost (4x 4 Gy + hyperthermia)
  Interventions: Radiation: Hypofractionated radiotherapy; Other: Hyperthermia

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — Preoperative hypofractionated 10x 3.25 Gy radiotherapy (5 consecutive days in a week, two weeks) prescribed on planned target volume (tumor volume + elective margins + setup/error margin) with daily image guidance with cone beam-CT or kV-portal position verification.
  Radiotherapy boost 4x 4 Gy within one week in case of unresectability after 6 weeks.
Other: Hyperthermia — Deep hyperthermia (Celsius TCS or BSD-2000) according to local protocol combined with radiotherapy, twice a week.

SUMMARY:
After a screening, which consists of biopsy, physical examination, initial diffusion-weighted magnetic resonance imaging (DWI-MRI) or body computed tomography (CT) scan, blood tests and case analysis on Multidisciplinary Team (MDT) meeting, a patient will receive the hypofractionated radiotherapy 10x 3.25 Gy with regional hyperthermia (twice a week) within two weeks. The response analysis in CT or DWI-MRI and toxicity assessment will be performed after at least 6 weeks. At the second MDT meeting, a final decision about resectability of the tumor will be made. In case of resectability or consent for amputation, if required, a patient will be referred to surgery. In case of unresectability or amputation refusal, the patient will receive the second part of the treatment which consists of 4x 4 Gy with hyperthermia (twice a week).

DETAILED DESCRIPTION:
There is a lack of standard treatment of unresectable and marginally resectable sarcomas. Results of commonly used approaches are unsatisfactory, especially in patients who are not candidates for neoadjuvant chemotherapy due to poor performance status, comorbidities, radioresistant pathology or disease progression on the commonly used chemotherapy regimens. The addition of regional hyperthermia to irradiation and in the prolonged gap between the end of hypofractionated 10x 3.25 Gy radiotherapy and surgery may allow obtaining the long-term local control with the maintenance of a good treatment tolerance.

Hypofractionation represents a variation of radiotherapy fractionation in which the total dose is divided into fewer fractions with an increased fraction dose. Such treatment may lead to additional biological effects when compared to conventionally fractionated radiotherapy (eg. vascular damage, increased immunogenicity, and antigenicity). The main advantages of hypofractionation are those related to the decreased overall treatment time which is more convenient for both patients and physicians, increased compliance and makes the treatment more cost-effective. Intriguing, such an approach may provide an additional benefit when treating non-radiosensitive tumors with a low alpha/beta ratio (eg. sarcomas).

Hyperthermia is a method of increasing the temperature in the tumor to damage cancer cells with minimum injury to the normal cells. It should be combined with another treatment modality (radio- or chemotherapy) rather than used alone. Its efficacy was proven in clinical trials. The treatment tolerance is usually very good.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent; age ≥18 years old
* Eastern Cooperative Oncology Group performance status 0 - 2
* Histologic diagnosis of locally advanced soft tissue sarcoma
* Marginally resectable or unresectable tumor (assessed at Multidisciplinary Tumor Board)
* Radioresistant sarcoma subtype (low-grade tumor or radioresistant histology) or contradictions to chemotherapy (assessed at Multidisciplinary Tumor Board) or progression after neoadjuvant chemotherapy

Exclusion Criteria:

* Radiation-induced sarcoma or previous radiation to the affected volume
* Histologic diagnosis of rhabdomyosarcoma (except pleomorphic subtype), osteogenic sarcoma, Ewing's sarcoma/PNET, aggressive fibromatosis
* Contraindications to radiotherapy or hyperthermia
* Distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the treatment schedule | Up to 3 months
  The exact 95% confidence interval for an estimated feasibility proportion of 80% (23 of 30 patients) does not include (60-80%) a value of 50%. Thus, for a sample size of 30 patients, the feasibility of 80% is above chance level performance (50%).

SECONDARY OUTCOMES:
One-year local control rate | 12 months after treatment completion
One-year progression-free survival | 12 months after treatment completion
One-year sarcoma-specific survival | 12 months after treatment completion
Rate of late toxicities | Two years after treatment completion
  Rate of late toxicities of a planned schedule of therapy according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Mateusz J Spałek, MD PhD, Principal Investigator — Maria Sklodowska-Curie National Research Institute of Oncology in Warsaw
Locations (1):
- Maria Sklodowska-Curie Institute - Oncology Center, Warsaw, Mazovian, Poland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication as supplementary materials
Time Frame: Data will be available since a publication (as a study supplementary material)
Access Criteria: Based on journal policy, open access is preferred

REFERENCES:
- [Background] Kosela-Paterczyk H, Szacht M, Morysinski T, Lugowska I, Dziewirski W, Falkowski S, Zdzienicki M, Pienkowski A, Szamotulska K, Switaj T, Rutkowski P. Preoperative hypofractionated radiotherapy in the treatment of localized soft tissue sarcomas. Eur J Surg Oncol. 2014 Dec;40(12):1641-7. doi: 10.1016/j.ejso.2014.05.016. Epub 2014 Sep 20. PMID 25282099
- [Background] Lindner LH, Issels RD. Hyperthermia in soft tissue sarcoma. Curr Treat Options Oncol. 2011 Mar;12(1):12-20. doi: 10.1007/s11864-011-0144-6. PMID 21360087
- [Background] Pennacchioli E, Fiore M, Gronchi A. Hyperthermia as an adjunctive treatment for soft-tissue sarcoma. Expert Rev Anticancer Ther. 2009 Feb;9(2):199-210. doi: 10.1586/14737140.9.2.199. PMID 19192958